CLINICAL TRIAL: NCT06985030
Title: Compliance of Head Positioning After Pars Planar Vitrectomy With Tamponade
Brief Title: Head Position Monitoring After Pars Planar Vitrectomy
Acronym: HPMPPV
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2404-050-1527
Record Dates: First submitted 2025-03-24; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Retinal Detachment; Macular Hole
MeSH Terms: conditions — Retinal Detachment; Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: gyroscope embedded eye-sheild — Small pcb with gyroscope and lithium polymer battery embedded eyeshield will be distributed right after surgery

SUMMARY:
In ophthalmic surgical practice, particularly for treating retinal detachment and macular hole disorders, vitrectomy procedures are routinely performed to remove the vitreous body followed by the injection of tamponade agents such as gaseous compounds (e.g., C3F8 or SF6) or silicone oil. These tamponade materials function by creating internal pressure against the retinal surface to facilitate reattachment. A critical determinant of surgical success in these cases is postoperative head positioning (prone posturing), as improper alignment may compromise the tamponade effect.

At the investigators' institution, participants undergoing such procedures are prescribed a strict prone position regimen for 7 consecutive postoperative days. This facedown positioning protocol aims to optimize interfacial contact between the tamponade agent and retinal tissue. However, conventional clinical practice faces a significant limitation: the inability to objectively verify patient compliance with prescribed postural guidelines outside clinical settings. Subjective patient reporting and intermittent clinical observations prove insufficient for quantifying adherence levels.

To address this critical gap in postoperative monitoring, the investigators propose implementing a novel electronic monitoring system integrated into therapeutic eye patches. This advanced device incorporates a miniaturized triaxial gyroscopic sensor array capable of continuously tracking cephalo-cervical orientation with high angular resolution. The system features complete electrical isolation from ocular tissues while maintaining sterility. Data acquisition occurs through a microSD card (capacity: 16GB) that logs positional parameters at 0.2Hz sampling frequency, creating comprehensive temporal records of head movement patterns.

ELIGIBILITY:
Inclusion Criteria:

* Patients who get vitrectomy

Exclusion Criteria:

* Patients who cannot maintain positioning due to their physical disability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who get vitrectomy with gas or silicone oil tamponade followed by positioning prescription
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
Compliance of head positioning | From enrollment to 7 days after surgery
  1. % time of right head positioning time (%)
  2. % time of applying eye patch time (%)
  3. Averaged deviation from instructed positioning (degree)
  4. % time of cotact between tamponade and retinal tear or macular hole (%)
  5. Questionaire (Visual Analogue Scale) :
     * pain, disability in daily life (dressing, eating, sleeping, washing, households)

SECONDARY OUTCOMES:
Baseline demographic and ocular characteristics | At enrollment
  1. Age (yr)
  2. Sex (male/female)
  3. Comorbities (if any), (ex. diabetes, hypertension, musculo-skeletal diseases)
  4. Baseline ocular characteristics
     * Visual acuity (logMAR)
     * Intraocular pressure (mmHg)
     * Wide fundus photo image
     * Optical Coherance Tomography image
     * Axial length (mm) (by ultrasonography A-scan, and IOL master)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, dep. of Ophthalmology, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided